CLINICAL TRIAL: NCT01049152
Title: Continuous Glucose Monitoring and Inflammation in Nondiabetic and Diabetic Patients Undergone Hemodialysis
Status: Completed | Type: Observational
Sponsor: University of Pavia (Other)
Responsible Party: Principal Investigator, Giuseppe Derosa, Professor, University of Pavia
Other Study IDs: 20090003173
Record Dates: First submitted 2010-01-12; First posted 2010-01-14 (Estimated); Last update posted 2022-05-24 (Actual); Status verified 2022-05

CONDITIONS: Diabetes; End Stage Renal Disease
Keywords: Diabetes mellitus; ESRD; CGM; Inflammation markers; Hemodialysis; Diabetic patients; Nondiabetic patients; All with ESRD; All undergone hemodialysis
MeSH Terms: conditions — Diabetes Mellitus; Kidney Failure, Chronic | interventions — Continuous Glucose Monitoring

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- nondiabetic patients: nondiabetic patients with ESRD undergone hemodialysis
  Interventions: Device: Continuous Glucose Monitoring (CGM)
- diabetic patients: diabetic patients with ESRD undergone hemodialysis
  Interventions: Device: Continuous Glucose Monitoring (CGM)

INTERVENTIONS:
Device: Continuous Glucose Monitoring (CGM) — CGM allocated one time for 3 days

SUMMARY:
Evaluation of different glycemic variations between the dialysis period and non-dialysis period in two groups: nondiabetic and diabetic patients undergone two different hemodialysis methods. Thirty-six patients, males and females, aged 50-80 years, with end stage renal disease (ESRD) will undergo hemodialysis and continuous glucose monitoring (CGM). The investigators will evaluate also inflammation markers before and after the different hemodialysis methods.

ELIGIBILITY:
Inclusion Criteria:

* patients with or without diabetes mellitus
* ESRD
* undergone hemodialysis
* males and females aged 50-80

Exclusion Criteria:

* tumors
* chronic inflammation diseases
* AMI
* acute pulmonary diseases

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: outpatients will undergo CGM at two different hemodialysis methods in a croos-over design. At the end of the study, it will evaluate inflammation markers intra-and inter-groups during the different hemodialysis methods.
Sampling Method: Non-Probability Sample
Enrollment: 36 (Actual)
Dates: Start 2009-07-31 (Actual); Primary Completion 2014-05-19 (Actual); Study Completion 2014-12-22 (Actual)

PRIMARY OUTCOMES:
-Hemodialysis tolerability -Hypoglycemia numbers -Hyperglycemia numbers -Inflammation markers | before and after each procedure

SECONDARY OUTCOMES:
variations of glycemia during the night; insulin-sensitivity | at the beginning of the first hemodialysis and at the end of the second hemodialysis

CONTACTS AND LOCATIONS:
Overall Officials: Giuseppe Derosa, MD, PhD, Principal Investigator — University of Pavia- Fondazione IRCCS Policlinico San Matteo
Locations (1):
- IRCCS Policlinico San Matteo, Pavia, Italy

REFERENCES:
- [Derived] Derosa G, Libetta C, Esposito P, Borettaz I, Tinelli C, D'angelo A, Maffioli P. Effects of two different dialytic treatments on inflammatory markers in people with end-stage renal disease with and without type 2 diabetes mellitus. Cytokine. 2017 Apr;92:75-79. doi: 10.1016/j.cyto.2016.12.026. Epub 2017 Jan 18. PMID 28110120
- [Derived] Derosa G, Libetta C, Esposito P, Borettaz I, Tinelli C, D'Angelo A, Maffioli P. Bicarbonate dialysis compared to hemodiafiltration on glycemic excursions in patients with end-stage renal disease with and without type 2 diabetes mellitus. J Diabetes Complications. 2015 Nov-Dec;29(8):1136-41. doi: 10.1016/j.jdiacomp.2015.08.009. Epub 2015 Aug 13. PMID 26387810